CLINICAL TRIAL: NCT06892860
Title: A Randomised Phase II Study Comparing 3 vs 6 Cycles of Platinum-based Chemotherapy Prior to Maintenance Avelumab in Advanced Urothelial Cancer
Brief Title: Comparing 3 vs 6 Cycles of Platinum-based Chemotherapy Prior to Maintenance Avelumab in Advanced Urothelial Cancer
Acronym: DISCUS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DISCUS
Record Dates: First submitted 2022-07-29; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Urinary Bladder Neoplasms
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 3 cycles of gemcitabine + cisplatin/carboplatin followed by avelumab (Experimental): Gemcitabine and cisplatin/carboplatin will be dispensed to patients on day 1 of each 21-day cycle of chemotherapy (3 cycles). Gemcitabine will additionally be dispensed to patients on day 8 of each 21-day cycle of chemotherapy. Following completion of gemcitabine and cisplatin/carboplatin chemotherapy, patients will then receive maintenance avelumab within 10 weeks of completing chemotherapy, on day 1 and 15 of each 28-day cycle for up to 2 years after the end of chemotherapy.
  Interventions: Drug: Avelumab
- 6 cycles of gemcitabine + cisplatin/carboplatin followed by avelumab (Active Comparator): Gemcitabine and cisplatin/carboplatin will be dispensed to patients on day 1 of each 21-day cycle of chemotherapy (6 cycles). Gemcitabine will additionally be dispensed to patients on day 8 of each 21-day cycle of chemotherapy. Following completion of gemcitabine and cisplatin/carboplatin chemotherapy, patients will then receive maintenance avelumab within 10 weeks of completing chemotherapy, on day 1 and 15 of each 28-day cycle for up to 2 years after the end of chemotherapy.
  Interventions: Drug: Avelumab

INTERVENTIONS:
Drug: Avelumab — Avelumab treatment will be given up to a maximum of 2 years from the end of chemotherapy

SUMMARY:
This is an adaptive, open-label, randomised phase II trial that aims to evaluate the impact of 3 vs 6 cycles of first-line platinum-based chemotherapy followed by maintenance avelumab in the quality of life of patients with locally advanced or metastatic urothelial cancer. Initially, 224 eligible and evaluable patients (112 in each arm) will receive 3 cycles vs 6 cycles of 3-weekly gemcitabine plus cisplatin/carboplatin, followed by 2-weekly maintenance avelumab until disease progression or intolerable toxicities. Avelumab treatment will be given up to a maximum of 2 years from the end of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent.
2. Ability to comply with the protocol, including but not limited to, the repeated completion of the EORTC QLQ-C30 questionnaires.
3. Age ≥ 18 years.
4. Histologically confirmed, unresectable locally advanced or metastatic urothelial carcinoma (i.e., cancer of the bladder, renal pelvis, ureter, or urethra). Patients with squamous or sarcomatoid differentiation or mixed cell types are eligible but a component of urothelial cancer is required.
5. Measurable disease by RECIST v1.1.
6. Eligible for gemcitabine/ cisplatin or gemcitabine/carboplatin. The following criteria are established for the use of carboplatin (patients not fulfilling the following carboplatin criteria should be considered for gemcitabine/ cisplatin):

   1. GFR <60 mL/min but ≥30 mL/min (measured by the Cockcroft-Gault formula or by local accepted standards). Subjects with a GFR ≥50 mL/min and no other cisplatin ineligibility criteria may be considered cisplatin-eligible based on the investigator's clinical judgement.
   2. ECOG or WHO performance status of 2.
   3. NCI CTCAE Grade ≥2 audiometric hearing loss.
   4. NYHA Class III heart failure.
7. Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0, 1 or 2.
8. Adequate haematologic and organ function as defined below:
9. Negative serum or urine pregnancy test within 2 weeks of Day 1 Cycle 1 for female patients of childbearing potential only.
10. Agreement to use adequate contraceptive measures

Exclusion Criteria:

* 1. Prior treatment with a PD-(L)-1 inhibitor for any advanced malignancy. Treatment with PD-(L)-1 inhibitors in the neoadjuvant or adjuvant setting for UC are permitted.

  2. Prior systemic therapy for locally advanced or metastatic urothelial carcinoma with the following exceptions: a platinum containing regimen (cisplatin or carboplatin) in the neoadjuvant or adjuvant setting if more than 6 months since last cycle have occurred. Patients who received adjuvant or neoadjuvant immune therapy for muscle invasive or non-muscle invasive disease are eligible.

  3. Pregnant and lactating female patients. 4. Known history of active CNS metastases. Patients with treated CNS metastases are permitted on the study if all of the following are true: 5. Prior allogeneic stem cell or solid organ transplantation. 6. Administration of a live, attenuated vaccine within 4 weeks prior to enrolment or anticipation that such a live, attenuated vaccine will be required during the study.

  7. Treatment with systemic immunostimulatory agents (including but not limited to interferons or interleukin [IL]-2) within 4 weeks or five half-lives of the drug, whichever is shorter, prior to enrolment (see section 11.26).

  8. Concurrent treatment with any other investigational agent or participation in another clinical trial with therapeutic intent within 4 weeks prior to enrolment.

  9. Evidence of significant uncontrolled concomitant disease that could affect compliance with the protocol or interpretation of results, including significant liver disease (such as cirrhosis, uncontrolled major seizure disorder, or superior vena cava syndrome).

  10. Malignancies other than urothelial carcinoma within 3 years prior to Cycle 1, Day 1, with the exception of those with a negligible risk of metastasis or death and treated with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, or ductal carcinoma in situ treated surgically with curative intent) or localized prostate cancer treated with curative intent and absence of prostate-specific antigen (PSA) relapse or incidental prostate cancer (Gleason score ≤ 3 + 4 and PSA < 10 ng/mL undergoing active surveillance and treatment naive). .

  11. Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or greater), myocardial infarction or cerebral vascular accident/stroke within 6 months prior to enrolment, unstable arrhythmias, or unstable angina.

  12. Radiotherapy within 2 weeks prior to C1D1. Patients must have recovered adequately from toxicities resulting from the intervention prior to starting study treatment.

  13. Major surgery (defined as requiring general anaesthesia and >24-hour inpatient hospitalization) within 4 weeks prior to randomisation. Patients must have recovered adequately from complications from the intervention prior to starting study treatment.

  14. History of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis on screening chest CT scan (History of radiation pneumonitis in the radiation field (fibrosis) is permitted).

  15. Active hepatitis infection (defined as having a positive hepatitis B surface antigen [HBsAg] test at screening) or hepatitis C. Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as having a negative HBsAg test and a positive antibody to hepatitis B core antigen [anti-HBc] antibody test) are eligible.

  16. Positive HIV test. 17. Active tuberculosis. 18. Active autoimmune disease including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis.

  19. History of autoimmune-related hypothyroidism, unless on a stable dose of thyroid replacement hormone.

  20. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies.

  21. Known hypersensitivity or allergy to biopharmaceuticals produced in Chinese hamster ovary cells or any component of avelumab.

  22. Active infection requiring systemic therapy. 23. Persisting toxicity related to prior therapy (NCI CTCAE Grade > 1); however, alopecia, sensory neuropathy Grade ≤ 2, or other Grade ≤ 2 not constituting a safety risk based on investigator's judgment are acceptable.

  24. Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results 25. Participants with previous or known history of allergic reaction to cisplatin, gemcitabine, carboplatin or other platinum containing compounds, or any component of the chemotherapy formulations.

  26. Patients with bleeding tumours 27. Any other contraindication for gemcitabine/ cisplatin or gemcitabine/carboplatin treatment as per SmPC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2021-12-16 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-22 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effect of 3 vs 6 cycles platinum-based, front-line chemotherapy followed by maintenance avelumab based on patient-reported outcomes (PROs) in the study population. | Cycle 6 (Arm A: 3x cycles of chemotherapy (21 days per cycle) plus 3x cycles of Avelumab (28 days per cycle), Arm B: 6 cycles of chemotherapy only (21 days per cycle)
  Change in GHS/QoL scale scores from baseline to completion of 6 cycles of treatment. Patients who withdraw from treatment between Cycles 4 and 6 will be included, provided an EORTC QLQ-C30 questionnaire is completed within 14 days from the date of withdrawal.

SECONDARY OUTCOMES:
To evaluate the effect of 3 vs 6 cycles platinum-based, front-line chemotherapy followed by maintenance avelumab based on additional patient-reported outcomes (PROs) in the study population. | 10 cycles of treatment (Arm A: 3x cycles of chemotherapy (21 days per cycle) plus 7x cycles of Avelumab (28 days per cycle), Arm B: 6 cycles of chemotherapy (21 days per cycle) followed by 4x cycles of avelumab (28 days per cycle))
  Quality of Life Assessment using the GHS/QOL scale score
To evaluate the effect of 3 vs 6 cycles platinum-based, front-line chemotherapy followed by maintenance avelumab based on clinician reported outcomes. | On completion of 6 cycles of treatment (From baseline to completion of cycle 6 (Arm A: 3x cycles of chemotherapy (21 days per cycle) plus 3x cycles of Avelumab (28 days per cycle), Arm B: 6 cycles of chemotherapy only (21 days per cycle)))
  Performance Status as measured by the Karnofsky Scale on completion of 6 cycles of treatment.
To evaluate the safety and tolerability of 3 vs 6 cycles of platinum-based, front-line chemotherapy followed by maintenance avelumab therapy. | From baseline throughout treatment (From baseline to completion of cycle 6 (Arm A: 3x cycles of chemotherapy followed by Avelumab, Arm B: 6 cycles of chemotherapy followed by Avelumab) for a maximum of 2 years on avelumab.
  Adverse events graded according to NCI-CTCAE v5.0
To assess the efficacy of 3 vs 6 cycles platinum based, front-line chemotherapy followed by maintenance avelumab in patients with advanced UC. | Baseline until end of trial participation (maximum of 2 years on avelumab)
  Efficacy endpoints

CONTACTS AND LOCATIONS:
Locations (3):
- Unicancer, Paris, France
- Adknoma, Madrid, Spain
- Barts Health NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Powles T, Hussain SA, Climent MA, Carbonero IG, Molina-Cerrillo J, Puente J, Borrega P, Malik J, Dourthe LM, Jones R, Castellano D, Duran I, Loriot Y, Priyadarshini G, Szabados B, Jamal F, Wang YQ, Kotriwala N, Jackson-Spence F, Ackerman C, Grande E. Three versus six cycles of platinum-based chemotherapy followed by avelumab maintenance as first-line treatment for advanced urothelial cancer: the phase II DISCUS trial. Ann Oncol. 2025 Oct 17:S0923-7534(25)04955-5. doi: 10.1016/j.annonc.2025.10.011. Online ahead of print. PMID 41110700